CLINICAL TRIAL: NCT01785576
Title: Couple-Based Intervention for Patients With Head and Neck Cancer and Their Partners
Acronym: CoupleCare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Rachel Pulido, Asst Director, Research Compliance, Endeavor Health
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: EH12-140
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Head and Neck Cancer
Keywords: couples; head and neck cancer; oncology; spousal support
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Couple-Based CBT Intervention (Experimental): Patients and partners will receive 4 sessions of a couple-based cognitive behavioral intervention focusing on communication and spousal support.
  Interventions: Behavioral: Couple-Based CBT Intervention
- Treatment as Usual (No Intervention): The treatment as usual group will complete all assessements and will not receive the psychosocial couple based intervention.

INTERVENTIONS:
Behavioral: Couple-Based CBT Intervention — Patients and partners will receive 4 sessions of a couple-based cognitive behavioral intervention focusing on communication and spousal support.
  Arms: Couple-Based CBT Intervention

SUMMARY:
The purpose of this study is to determine whether a brief couple-based supportive intervention effectively assists patients and their partners coping with the challenges of head and neck cancer.

DETAILED DESCRIPTION:
This intervention will adapt a well-validated cognitive-behavioral therapeutic approach in a four-session intervention to teach patients and partners specific couple-based cancer-focused support skills. In addition, in order to gather information on outcome variables, couples will complete three assessments during the course of treatment (pre-treatment, following treatment, and six month follow-up). These assessments will include questionnaire measures as well as couple communication whereby couples will participate in two videotaped conversations whereby one partner of the couple discusses a concern and the other member of the couple provides support. We also will implement a "daily diary" assessment whereby day-to-day psychological and physical symptoms experienced by the patient and partner will be assessed and daily effects of the intervention can be analyzed. Patients and partners will participate in the daily diary portion of the study following the post-assessment. They will be emailed an electronic link to a brief questionnaire daily for 7 days. The items in this daily assessment will comprise questions that are part of the general assessment measures such as dyadic coping, spousal support, and relationship satisfaction. The patient will also complete questions about pain and fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Recently diagnosed with Head and Neck Cancer receiving chemotherapy and/or radiation therapy
* No history of cancer within past 3 years (other than basal cell)
* Living with partner in a committed relationship at least 6 months
* Patient and partner speak and read English

Exclusion Criteria:

* Serious cognitive or emotional issues that preclude full participation in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Quality of Life | 6 months

SECONDARY OUTCOMES:
Spousal Support | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tina Gremore, PhD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States

REFERENCES:
- [Derived] Gremore TM, Brockstein B, Porter LS, Brenner S, Benfield T, Baucom DH, Sher TG, Atkins D. Couple-based communication intervention for head and neck cancer: a randomized pilot trial. Support Care Cancer. 2021 Jun;29(6):3267-3275. doi: 10.1007/s00520-020-05848-5. Epub 2020 Oct 26. PMID 33106976